CLINICAL TRIAL: NCT02774681
Title: A Phase II Single Arm Study of Palbociclib in Patients With Metastatic HER2-positive Breast Cancer With Brain Metastasis
Brief Title: Palbociclib in Treating Patients With Metastatic HER-2 Positive Breast Cancer With Brain Metastasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Northwestern University (Other)
Collaborators: Pfizer (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 15B08; STU00202582 (CTRP (Clinical Trial Reporting Program)); NU 15B08 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-00626 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Breast Carcinoma Metastatic in the Brain; Estrogen Receptor Negative; HER2/Neu Negative; HER2/Neu Positive; Progesterone Receptor Negative; Recurrent Breast Carcinoma; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mental Status and Dementia Tests; palbociclib; Trastuzumab; PF-05280014

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (palbociclib) (Experimental): Patients receive palbociclib PO daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with HER2 positive breast cancer may also receive trastuzumab IV over 30-90 minutes every 3 weeks.
  Interventions: Procedure: Cognitive Assessment; Drug: Palbociclib; Procedure: Quality-of-Life Assessment; Biological: Trastuzumab

INTERVENTIONS:
Procedure: Cognitive Assessment — Ancillary studies
Drug: Palbociclib — Given PO
  Other Names: Ibrance; PD-0332991; PD-332991
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; PF-05280014; rhuMAb HER2; RO0452317; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar PF-05280014

SUMMARY:
The purpose of this study is to evaluate if the study drug palbociclib has anti-tumor activity against the breast cancer that has spread to the brain and also to determine the overall radiographic response rate in the CNS. Palbociclib is an anti-cancer medication that has been shown to stop cancer cells from growing. It has been approved in hormone positive breast cancer, along with other hormone therapies and has been found to be effective. The preclinical studies suggest that the drug may also have activity in other types of breast cancer, such as HER2 positive breast cancer. The purpose of this study is to see if the study drug is effective in patients with brain metastasis, who have HER2-positive breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the radiographic response rate in the central nervous system (CNS) in patients with HER2-positive breast cancer who have brain metastasis treated with palbociclib.

SECONDARY OBJECTIVES:

I. To determine the progression-free survival (PFS) and overall survival (OS) in patients with HER2-positive breast cancer who have brain metastasis treated with palbociclib.

II. To determine time to CNS progression in patients with HER2-positive breast cancer who have brain metastasis treated with palbociclib.

III. To determine systemic overall response rate (ORR) in patients with HER2-positive breast cancer who have brain metastasis treated with palbociclib.

IV. To determine the safety and tolerability of palbociclib in patients with and HER2-positive breast cancer.

TERTIARY OBJECTIVES:

I. To evaluate circulating tumor deoxyribonucleic acid (DNA) at baseline, 2 month and 4 months; particularly to assess cyclin D1 aberrations, and if this is predictive of responses.

II. To evaluate genomic landscape of available CNS and non-CNS tumors, and describe any discordance.

III. To evaluate cognitive function and quality of life at baseline, 2 and 4 months in patients receiving palbociclib.

OUTLINE:

Patients receive palbociclib orally (PO) daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with HER2 positive breast cancer may also receive trastuzumab intravenously (IV) as standard of care concurrently with palbociclib.

After completion of study treatment, patients are followed up at 3, 6, 9, and 12 months, and then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HER2-positive metastatic breast cancer (estrogen and progesterone receptor 0%, HER-2 3+ by immunohistochemistry (IHC); if IHC score of 2, fluorescence in situ hybridization (FISH) ratio must be greater than 2.0; if FISH less than 2.0, HER2 copy number must be greater than 6; NOTE: Brain lesions are not required to have pathologic confirmation
* Patients should not have received > 2 lines of chemotherapy for metastatic disease
* Patients must have a life expectancy of at least 12 weeks at the time of registration
* Eastern Cooperative Oncology Group (ECOG) performance status >= 2
* Measurable disease in the brain, defined as at least 1 lesion measuring >= 5 mm on imaging at the time of registration
* If patients are on corticosteroids, they must have been on a stable or decreasing dose >= 5 days prior to obtaining their baseline gadolinium (Gd)-magnetic resonance imaging (MRI) of brain; this MRI is to be obtained within 28 days of registration; NOTE: If patient needs escalation of steroids prior to therapy, or are on unstable doses of steroids they are not eligible
* Patients who underwent neurosurgery (NSGY) or stereotactic radiosurgery (SRS) to a brain lesion must have a new measureable lesion; NOTE: SRS may be done to a lesion that will not be used for response evaluation and should be done > 2 weeks prior to registration; any NSGY procedure must have been completed > 3 weeks prior to registration
* Patients must not have received systemic therapy within 2 weeks of initiating palbociclib; NOTE: For the HER2-positive cohort, patients on trastuzumab can remain on the drug; no break or washout period required; however, lapatinib, ado-trastuzumab-emtansine, and pertuzumab are prohibited and a minimum wash out period of 2 weeks is required
* Patients must exhibit adequate bone marrow, liver, and renal function, within 14 days prior to registration, defined as:

  * Absolute neutrophil count (ANC) >= 1,000/mm^3 (growth factor support is permitted)
  * Platelets >= 100,000/mm^3 (may be reached by transfusion)
  * Hemoglobin >= 10 gm/dl (may be reached by transfusion)
  * Glutamate pyruvate transaminase (GPT)/glutamate oxaloacetate transaminase (GOT) < 3 x upper limit of normal (ULN) (or < 5 x ULN in case of liver metastasis)
  * Bilirubin < 3 x ULN (or < 5 x ULN in case of liver metastasis)
  * Creatinine < 1.5 x ULN
* Females of child-bearing potential (FOCBP) and males must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 2 weeks following completion of therapy; should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; likewise, if the female partner of a male patient becomes pregnant while participating in this study, he should inform his treating physician immediately; NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy
  * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* Female patients must have a negative urine pregnancy test within 7 days prior to registration; if urine test is positive, it should be followed by serum pregnancy test
* Patients must sign an informed consent prior to registration and before undergoing any study-specific procedures indicating that they are aware of the investigational nature of this study
* Patient must have the ability to swallow and retain oral medication
* Patient must have the ability to comply with all study requirements

Exclusion Criteria:

* Any uncontrolled neurological symptom attributed to CNS metastasis
* Brain metastasis must not be impending herniation or other significant vasogenic edema requiring increasing steroid doses; lesions must not have frank hemorrhage
* Patients with leptomeningeal disease are not eligible for participation
* Any significant medical illnesses or infection that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy are not eligible for participation
* Known human immunodeficiency virus (HIV) positive status
* Known active hepatitis B and/or C
* Previous treatment with palbociclib
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to palbociclib are not eligible; AND/OR patients who have had prior exposure to compounds of similar chemical or biologic composition to palbociclib are not eligible hypersensitivity to any component of palbociclib are not eligible for participation
* Patients being treated with any other experimental agents/clinical trials are not eligible for participation; if the patient is on any investigational agent, a wash-out period of minimum 2 weeks prior to registration is mandatory for the patient to be eligible for the study
* Patients who are on any prohibited medication; a wash-out period of minimum 2 weeks prior to registration is mandatory for the patient to be eligible for the study
* Inability to swallow capsules, malabsorption syndrome or gastrointestinal disease that severely affects the absorption of study drugs, major resection of the stomach or small bowel, or gastric bypass procedure
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Ongoing or active infection requiring systemic treatment
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia: except atrial fibrillation (AF) and supraventricular tachycardia (SVT) that are controlled by medication
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Female patients who are pregnant or nursing are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2020-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristofanilli Massimo, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Northwestern Lake Forest Hospital, Lake Forest, Illinois
  - Houston Methodist Hospital/Houston Methodist Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual May 25, 2016 with the first patient being treated on study August 31,2016. the total accrual goal of 25 patients. The study closed to further accrual January 28, 2019 with 12 patients enrolled on the study
Period: Treatment on Study
Arm/Group | Treatment (Palbociclib)
Started | 12
Reached 1st Response/2 Cycles | 10
Went on to Start Cycle 3 | 5
Completed | 5
Not Completed | 7
Not completed — Progressive Disease | 7
Period: Follow-Up for 3 Years
Arm/Group | Treatment (Palbociclib)
Started | 12
Completed | 0
Not Completed | 12
Not completed — Death | 11
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 55 [44 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Response Rate (RRR) in the CNS in Patients With HER2-positive Breast Cancer Who Have Brain Metastasis Treated With Palbociclib
Description: Assess the Radiographic Response Rate (RRR) in the CNS by modified Response Assessment in Neuro-Oncology Criteria Brain Metastasis (modifiedRANO-BM). Maximum response prior to disease progression will be used. In General:
  Complete Response : Disappearance of all lesions Partial Response: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
  Progressive Disease: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression.)
Time Frame: Up to 3 years
Population: Below table shows best response (Clinical and radiological) of all patients treated on study. Patients that did not complete 2 cycles of treatment required for evaluability for response rate objective are shown. No RRR was not calculated as the study did not met statistical analysis criteria due to study closing before total accrual was met.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 12
Participants
  Stable Disease CNS | 6
  Progressive Disease CNS | 6

2. Secondary Outcome: Incidence of Adverse Events
Description: Determine the safety and tolerability of palbociclib in patients with HER2-positive breast cancer by evaluating number, frequency, and severity of adverse events using Common Terminology Criteria for Adverse Events version 4.03. The number of patients that experienced SAEs that were determined to be at least possibly related to study drug are reported below.
Time Frame: Up to 3 years
Population: Data not collected for analysis
Measure: Number; unit: participants
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 12
participants | 1

3. Secondary Outcome: Overall Survival (OS)
Description: Evaluate OS in patients with HER2-positive breast cancer who have brain metastasis treated with palbociclib. OS is defined as the time from treatment initiation until death due to any cause. Number of patients remaining alive as of the last follow up date, is reported below.
Time Frame: Up to 3 years
Population: one patient withdrew consent to be followed for survival
Measure: Number; unit: participants alive
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 11
participants alive | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Determine the PFS in patients with HER2-positive breast cancer who have brain metastasis treated with palbociclib where PFS is defined as the time from treatment initiation to documented disease progression or death for any reason. Below shows the number of patient who discontinued treatment due to progression of disease.
Time Frame: Up to 3 years
Population: Not sufficient patients enrolled for statistical analysis due to study closing to accrual before the accrual goal was met. Number of patients shown below is the number of patients that discontinued treatment due to progression.
Measure: Number; unit: patients
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 12
patients | 11

5. Secondary Outcome: Overall Response Rate (ORR)
Description: Evaluate systemic ORR defined as partial response or complete response assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 where:
  Complete Response = complete disappearance of all lesions Partial Response = At least 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to 3 years
Population: All patient data is shown. Patients that did not complete 2 cycles of treatment required for response are also included as there was no analysis of the data.
Measure: Number; unit: participants
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 12
participants | 0

6. Secondary Outcome: Time to CNS Progression
Description: Time to CNS progression will be defined as the time from treatment initiation to documented disease progression (modified RANO-BM criteria) in the CNS.
Time Frame: Up to 3 years
Population: Data not collected. Not sufficient patients enrolled for statistical analysis due to study closing to accrual before the accrual goal was met.
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Change in Cognitive Function in Patients Receiving Palbociclib
Description: Change in cognitive function will be assessed at baseline, 2 months and 4 months and will be collected using patient reported outcome questionnaires: Functional assessment of Cancer Therapy-Cognitive function Version 3.0 (Fact -Cog)
Time Frame: At baseline, 2 months and 4 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Genomic Landscape of Available CNS and Non-CNS Tumors
Description: To evaluate genomic landscape of available CNS and non-CNS tumors, and describe any discordance. Genotyping of CNS and non-CNS tumors will be performed from archival tissue that will be obtained at baseline. Genotyping will be performed through commercial next generation sequencing assays.
Time Frame: At baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Quality of Life in Patients Receiving Palbociclib
Description: Quality of life measures will be assessed at baseline, 2 months and 4 and will be collected using patient reported outcome questionnaires: Functional Assessment of Cancer Therapy-Brain (FACT-Br) Version 4.0
Time Frame: At baseline, 2 months and 4 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Cyclin D1 Aberrations Assessed by Circulating Tumor DNA
Description: Analyze circulating tumor DNA to assess cyclin D1 aberrations and if this is predictive of response to treatment. Circulating tumor DNA will be collected from whole blood at baseline, 2 and 4 months through commercial next generation sequencing assays.
Time Frame: At baseline, 2 months and 4 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over a 2 and half year period for the study. For each patient they were collected from treatment initiation until 30 days post the last treatment with range of cycles completed by patients being less than 1 Cycle to 5 Cycles (1 Cycle = 28 Days)
Arm/Group | Treatment (Palbociclib)
All-Cause Mortality (participants affected / at risk) | 11/12
Serious Adverse Events (participants affected / at risk) | 6/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Palbociclib) (N=12)
Confusion (Psychiatric disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 2 (2)
Seizure (Nervous system disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Palbociclib) (N=12)
Anemia (Blood and lymphatic system disorders) | 8
Hypothyroidism (Endocrine disorders) | 1
Blurred Vision (Eye disorders) | 1
Watery Eyes (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Stomach Pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 5
Flu Like Symptoms (General disorders) | 1
Gait Disturbance (General disorders) | 2
Malaise (General disorders) | 1
Pain (General disorders) | 2
Tooth Infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 4
Creatinine Increased (Investigations) | 2
Lymphocyte Count Decreased (Investigations) | 7
Neutrophil Count Decreased (Investigations) | 8
Platelet count Decreased (Investigations) | 6
White Blood Cell Decreased (Investigations) | 10
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Memory Impairment (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Chronic Kidney Disease (Renal and urinary disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 1
Low GFR (Investigations) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Stomatitis (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study was closed before the accrual goal was met due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT02774681/Prot_SAP_000.pdf